CLINICAL TRIAL: NCT05874024
Title: Induction of Labour With a Double Balloon Catheter - Comparison of Effectiveness of Six Versus Twelve Hours Placement: a Prospective Case Control Study
Brief Title: Induction of Labour With a Double Balloon Catheter
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DBK-Trial
Record Dates: First submitted 2023-04-13; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Labor, Induced
Keywords: double balloon catheter; cervical ripening; time to delivery
MeSH Terms: interventions — Labor, Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Placement 6 hours: double balloon catheter placement for 6 hours
  Interventions: Procedure: induction of labour with double balloon catheter placement for 6 hours
- Placement 12 hours: double balloon catheter placement for 12 hours
  Interventions: Procedure: induction of labour with double balloon catheter placement for 12 hours

INTERVENTIONS:
Procedure: induction of labour with double balloon catheter placement for 6 hours — catheter placement for 6 hours beginning in the morning at around 8 a.m.
  Groups: Placement 6 hours
Procedure: induction of labour with double balloon catheter placement for 12 hours — catheter placement for 12 hours in the evening at around 8 p.m.
  Groups: Placement 12 hours

SUMMARY:
The objective of this study is to provide a comprehensive analysis of various time intervals (1:1). In addition to evaluating the time interval until delivery after completion of induction, the study also aims to investigate the rate of vaginal births and the type of combination therapy used (including the method of implementation and subsequent induction).

DETAILED DESCRIPTION:
Approximately 22% of births in Germany are induced annually using either medicinal, mechanical, or sequential mechanical/medicinal methods, with oxytocin and prostaglandins being the available drug options. Double balloon catheters have been used in clinics for over a decade for mechanical induction of labour, resulting in cervical ripening and possible onset of labour through endogenous prostaglandin release. This method is associated with low rates of uterine tachysystole and maternal and neonatal morbidity.

The recommended placement time for the double balloon catheter is 12 hours, typically performed at night in an inpatient setting, which may cause early exhaustion and fatigue for patients. However, a study has shown that a shorter insertion time of 6 hours is equally safe and effective, without any time savings beyond the shortened insertion time.

This study aims to investigate the feasibility and effectiveness of shortening the induction birth interval from 12 to 6 hours. The investigators hypothesize that this will result in a shorter induction birth interval with comparable maternal and neonatal outcomes. This analysis will test the effectiveness of the shortened induction birth interval.

ELIGIBILITY:
Inclusion Criteria:

* destational age above or equal 37/0 weeks of gestation
* desired spontanous delivery
* Bishop-Score below or equal to 5
* cranial position
* single pregnancy

Exclusion Criteria:

* unable to consent
* pathological CTG according FIGO criteria

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: tertiary center, women undergoing induction of labour
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
induction to delivery interval | From date and time of beginning of labour induction to date and time of birth, assessed as long as needed, but not longer than 5 days
  the induction to delivery interval measured in minutes

SECONDARY OUTCOMES:
number of participants with sequential drug induction of labour | assessd after double balloon catheter placement until time of birth, but not longer than 3 days
  the need for additional drugs for inductionof labour after the assigned placement time of the double balloon catheter
prostaglandin to delivery interval | From date and time of beginning of prostaglandin treatment to date and time of birth, assessed as long as needed, but not longer than 3 days
  the prostaglandin to delivery interval measured in minutes
mode of delivery | after induction of labour at time of delivery
  resulting mode of delivery after induction of labour expressed as spontaneous vaginal, vaginal operative or caesarean section
blood loss during delivery | at time of delivery
  maternal outcome blood loss during delivery in ml
number of participants with uterine rupture | at time of delivery
  maternal outcome uterine rupture
arterial umbilical pH | at time of delivery
  neonatal outcome arterial umbilical pH measured directly after delivery
arterial umbilical base excess | at time of delivery
  neonatal outcome arterial umbilical base excess measured directly after delivery
number of participants neonatal acidosis | at time of delivery
  neonatal outcome arterial umbilical pH < 7.1
apgar 5 min | 5 minutes after delivery
  neonatal outcome apgar 5 min (A- appearance, P-Pulse, G- grimace, A- activity, R-respiration) with a range between 0-10 with higher values as better outcome
number of participants with pathological cardiotocography (CTG) | at time of labour induction
  neonatal outcome pathological CTG (cardiotocography) at time of labour induction
number of participants with meconium-containing amniotic fluid | at time of delivery
  neonatal outcome meconium-containing amniotic fluid measured as visible green stained amniotic fluid at time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Schleußner, Prof. Dr., Principal Investigator — Jena University Hospital, Department of Obstetrics
Locations (1):
- Jena University Hospital, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No